CLINICAL TRIAL: NCT06280664
Title: Efficacy Of Hiatal Closure For GERD
Status: Recruiting | Type: Observational
Sponsor: University of Chicago (Other)
Responsible Party: Sponsor
Other Study IDs: IRB20-1151
Record Dates: First submitted 2024-02-19; First posted 2024-02-28 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2026-01

CONDITIONS: Gastro Esophageal Reflux
MeSH Terms: conditions — Gastroesophageal Reflux

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The purpose of this protocol is to study the efficacy of hiatal closure for early GERD disease. The study team hypothesizes that hiatal closure for early GERD disease is an efficacious treatment of GERD.

DETAILED DESCRIPTION:
Gastro-Esophageal Reflux Disease (GERD) affects 60 million Americans involving an estimated 20 million Americans dependent on long term medication to control symptoms and progression of the disease. Although surgical hiatal hernia repair and creation of an anti-reflux valve can correct the underlying cause of GERD by repairing the anatomic defect and reestablishing the competency of the lower esophageal sphincter (LES), only 24,000 patients annually undergo surgery for GERD. However, with the advent of minimally invasive laparoscopic techniques to treat GERD, more patients at early phases of the disorder are being surgically treated.

The traditional approach to surgical treatment of GERD has been hiatal hernia repair with Nissen fundoplication. However, fundoplication itself may be unnecessary for recovery of the lower esophageal sphincter. Several groups have demonstrated that partial or even minimal wrapping of the esophagus achieves equal control of GERD to complete wrapping. Despite extensive geometric and physics-based explanations for this observational enigma, the science underlying these highly reproducible observations across surgeons and continents remains poorly understood. Furthermore, outcomes following hiatal hernia repair alone for the treatment of GERD have not been studied since before the advances in laparoscopic technique.

Because of the high-volume gastrointestinal surgery center, the study team has the opportunity to rigorously study patient-centered outcomes and the disease processes as they are treated with this surgery. These outcomes after hiatal closure alone have not been published with the use of minimally invasive techniques where rigorous repairs can be achieved and thus, the study team is seeking this opportunity to demonstrate the efficacy of hiatal closure alone and recovery of the lower esophageal sphincter in those patients with symptomatic GERD and small hiatal defects. Publishing outcomes of this technique would represent a great leap forward in enhancing the knowledge base upon which to define the principles and techniques for the surgical treatment of GERD.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 - 50 years
* Able to provide informed consent
* BMI <30
* Hiatal defect <4cm on esophagram
* pH testing requirement: pH <4 for >5.5%
* Surgical candidate for hiatal closure only

Exclusion Criteria:

* Vulnerable subjects (children, prisoners, pregnant women) will be excluded.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: The estimated annual number of subjects enrolled prospectively in the study is 20. The recruitment goal is 40. The research team will screen all patients that are being followed-up at the gastrointestinal surgery clinic at the UCM.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2020-10-02 (Actual); Primary Completion 2028-10 (Estimated); Study Completion 2028-10 (Estimated)

PRIMARY OUTCOMES:
Concentration of pH testing | at 1 and 2 years
  Determine GERD remission for hiatal closure alone for patients with pH proven GERD

CONTACTS AND LOCATIONS:
Overall Officials: Yalini Vigneswaran, MD, Principal Investigator — University of Chicago
Locations (1):
- The University of Chicago, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No